CLINICAL TRIAL: NCT06582290
Title: Investigating the Clinical Utility of the Oxford Virtual Autism Assessment Tool (OVAAT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Health NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: OxfordNHS
Record Dates: First submitted 2024-08-28; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder; Healthy; Neurotypical
Keywords: Autism Spectrum Disorder; ASD; OVAAT; Evaluation; Clinical utility
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The study will use a correlational design. An online autism assessment tool (the Oxford Virtual Autism Assessment Tool (OVAAT)) will be (a) compared to an existing standardised autism observation tool (the ADOS-2) and developmental history (gathered from parents) in terms of it's ability to identify features of ASD and (b) evaluated to determine whether it can distinguish between 13-18 year old young people with ASD and 13-18 year old young people with no neurodevelopmental conditions or mental health problems.
Who Masked: Outcomes Assessor
Masking Description: The two clinicians completing and coding the OVAATs will be blind to which group the participant is.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autistic (Experimental): This will be participants who are waiting for an autism assessment in the Oxfordshire CAMHS Neurodevelopmental Conditions (NDC) pathway. The participant are will complete the OVAAT and an ADOS-2 assessment.
  The participant will have a neurodevelopmental assessment using the ADOS-2 is an existing tool that we use to assess autism and a developmental history - this is the current standard assessment process. They will receive feedback from this appointment. The second appointment will be using the OVAAT. This assessment will be video and audio recorded (through Microsoft Teams) so that we can check whether another clinical researcher comes to the same conclusion as the person providing the OVAAT. We will only keep the recording until the 2nd researcher has watched and listened to the recording.
  Interventions: Diagnostic Test: Oxford Virtual Autism Assessment Tool (OVAAT)
- Neurotypical (Experimental): These participants will be neurotypical young people recruited from the general population of Oxfordshire. They will only receive an OVAAT appointment.
  The participants will first complete screening measures to assess their eligibility for the study. If they are still eligible, an OVAAT appointment will be arranged. This will be the same process as group 1. This assessment will be video and audio recorded (through Microsoft Teams) so that we can check whether another clinical researcher comes to the same conclusion as the person providing the OVAAT. We will only keep the recording until the 2nd researcher has watched and listened to the recording.
  Interventions: Diagnostic Test: Oxford Virtual Autism Assessment Tool (OVAAT)

INTERVENTIONS:
Diagnostic Test: Oxford Virtual Autism Assessment Tool (OVAAT) — The OVAAT is an online ASD diagnostic tool that has been designed to identify both the external/observable features of autism but also the internal/experiential features of autism.

SUMMARY:
The goal of the study is to evaluate a new Autism Spectrum Disorder (ASD) diagnostic tool (Oxford Virtual Autism Assessment Tool (OVAAT)) to see whether it can:

* Be able to identify autistic traits
* Be able to distinguish between autistic and non-autistic young people
* Is the tool better, similar or worse than another evidence-based observational tool (ADOS-2) in identifying features of autism?

DETAILED DESCRIPTION:
Background and study aims:

Standardised tools (i.e. tools that have been formally researched/evaluated) are a key part of ASD assessments. Some young people prefer online to face-to-face assessments. Recent research indicates that some young people with ASD show fewer observable features/symptoms of ASD but describe internal features/symptoms of ASD. At present, there is (a) no standardised virtual/online assessment tool and (b) no standardised tool which balances gathering information about observable features of ASD and self-reported features of ASD. This study will begin the process of scientifically evaluating the OVAAT (a video-based tool assessing both observable and self-reported features of ASD).

Who can participate? The study will have two groups: group 1 will be 13-18 year old young people waiting for an autism assessment in the Oxfordshire CAMHS Neurodevelopmental Conditions (NDC) pathway who have access to and are able to use a laptop or desktop computer and a quiet place to complete the assessment. Group 2 will be 13-18 year old young people with no neurodevelopmental or mental health conditions who have access to and are able to use a laptop or desktop computer and a quiet place to complete the assessment.

What does the study involve? Group 1: Participants will complete the OVAAT and an ADOS-2 assessment. The OVAAT is the tool that is being tested. The ADOS-2 is an existing tool that is used to assess autism and participants would complete this as part of the standard assessment. The OVAAT assessment will be video and audio recorded (through Microsoft Teams) so that the investigators can check whether another clinical researcher comes to the same conclusion as the person providing the OVAAT. The investigators will only keep the recording until the second researcher has watched and listened to the recording.

Group 2: Participants will complete some questionnaires that identify potential features of autism, ADHD and common mental health problems. Participants will also meet with a clinical researcher from the NDC team to complete the OVAAT. The OVAAT assessment will be video and audio recorded (through Microsoft Teams) so that the investigators can check whether another clinical researcher comes to the same conclusion as the person providing the OVAAT. The recordings will only be kept until the second researcher has watched and listened to the recording.

What are the possible benefits of participating? Participants will be given a £10 Amazon voucher for taking part (for group 2, participants will need to complete the screening measures (participants must pass the screening) and the OVAAT before receiving the voucher. For group 1, participants will need to complete the diagnostic assessment and the OVAAT before receiving the voucher). The investigators also hope that this study will help to determine whether this new tool (the OVAAT) is better than existing tools at identifying autism and give young people a better experience during their assessment.

What are the possible risks of participating? There are no significant risks to taking part. However, the questionnaires or OVAAT could identify potential neurodevelopmental features or symptoms of mental health problems. If this happens, participants and/or their parents will be given information about how to access further support.

It is possible that participants confidentiality might need to be broken (e.g. if there is a risk of significant harm to the participant or others). If this is the case, every effort will be made to discuss this with the participant (unless this would e.g. increase the risk of harm). If there is a significant risk of harm to the participant or someone else, only people who need to be informed of the risk (i.e. those who can mitigate the risk and prevent harm) will be informed (e.g. GP, emergency services, CAMHS professionals, parents/caregivers) and they will only be provided with information relevant to the risk. Participants (and their parents/caregivers, where appropriate) will be informed of what information has been shared, and with whom.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: 13-18 year old young people waiting for an autism assessment in the Oxfordshire CAMHS Neurodevelopmental Conditions (NDC) pathway who have access to and are able to use a laptop or desktop computer and a quiet place to complete the assessment.
* Group 2: 13-18 year old young people with no neurodevelopmental or mental health conditions who have access to and are able to use a laptop or desktop computer and a quiet place to complete the assessment.

Exclusion Criteria:

* Group 1: 13-18 year old young people waiting for an autism assessment in the Oxfordshire CAMHS NDC pathway who have an existing or suspected neurodevelopmental diagnosis other than autism (e.g. ADHD, Learning Disability) or significant mental health problem (e.g. major depression, psychosis, eating disorder) and/or who are unable to speak English fluently.
* Group 2: 13-18 year olds with any suspected or current neurodevelopmental or mental health conditions and/or who are unable to speak English fluently.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Oxford Virtual Autism Assessment Tool (OVAAT) | Up to 3 weeks after recruitment
  The OVAAT is an online ASD diagnostic tool that has been designed to identify both the external/observable features of autism but also the internal/experiential features of autism.

SECONDARY OUTCOMES:
Revised Children's Anxiety and Depression Scale (and Subscales) (RCADS) | Day 0
  Used in the screening for group 2 47 item questionnaire scored on a scale of 0-3, with 0 being "never" and 3 being "always"). Participants in group 2 will score statements based on how often the things (statements) happen to them e.g., "I worry about things".
Autism Spectrum Quotient (AQ-10) | Day 0
  Used in group 2 screening process. 10 item measure that looks at whether a person should be be referred for further autism assessment. Participants are asked to indicate their level of agreement on 10 statements (on a scale of 1-4, 1 being "definitely agree" to 4 "definitely disagree").
Adult ADHD Self-Report Scale (ASRS) | Day 0
  Used in the group 2 screening process 18-item questionnaire spilt into 2 parts (part a. and part b.). Participants are asked to score rate themselves based on how they have felt and conducted themselves over the past six months (using "never", "rarely", "sometimes", "often" or "very often").
Prodromal Questionnaire (PQ-16) | Day 0
  Used in group 2 screening process. 16-item questionnaire that asks participants to either indicate "true" or "false" for 16 items that look at the risk of potential psychosis. For any statements that participants indicate as "true" they are asked to rate their level of distress (on a scale of 0-3, with 0 being "none" and 3 being "severe").
Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) | Within 2 to 3 months of consent form being signed
  This used before the OVAAT and is used in the diagnostic assessment in group 1. The ADOS-2 is an observation-based tool used to assess and diagnose ASD. It uses a combination of questions and activities to assess and evaluate a person's communication skills, social interaction and imaginative se of materials.

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Health NHS Foundation Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the participants age and because the IPD may contain identifiable or sensitive information it is unlikely this will be shared outside of the trust.

REFERENCES:
- [Background] Schutte JL, McCue MP, Parmanto B, McGonigle J, Handen B, Lewis A, Pulantara IW, Saptono A. Usability and reliability of a remotely administered adult autism assessment, the autism diagnostic observation schedule (ADOS) module 4. Telemed J E Health. 2015 Mar;21(3):176-84. doi: 10.1089/tmj.2014.0011. Epub 2015 Jan 8. PMID 25569603

DOCUMENTS (1):
  • Informed Consent Form (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT06582290/ICF_000.pdf